CLINICAL TRIAL: NCT01107457
Title: A Dose-Ranging And Efficacy Study of LY2439821 (An Anti-IL-17 Antibody) In Patients With Moderate-To-Severe Psoriasis
Brief Title: A Study in Participants With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12060; I1F-MC-RHAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-14; First posted 2010-04-21 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis
Keywords: Moderate; Severe; Plaque; Chronic
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular; Plaque, Amyloid; Bronchiolitis Obliterans Syndrome | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 10 mg Ixekizumab (Experimental): Part A:
  10 milligrams (mg) ixekizumab given subcutaneous (SC) on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through approximately week 344.
  Interventions: Biological: Ixekizumab
- 25 mg Ixekizumab (Experimental): Part A:
  25 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC (Q4W). Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through approximately week 344.
  Interventions: Biological: Ixekizumab
- 75 mg Ixekizumab (Experimental): Part A:
  75 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through approximately week 344.
  Interventions: Biological: Ixekizumab
- 150 mg Ixekizumab (Experimental): Part A:
  150 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  Administered 120 mg ixekizumab SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional) 80 mg ixekizumab given SC Q4W through approximately week 344.
  Interventions: Biological: Ixekizumab
- Placebo (Placebo Comparator): Part A:
  Placebo given on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional) 120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through approximately week 344.
  Interventions: Biological: Ixekizumab; Drug: Placebo
- 120 mg Ixekizumab (Experimental): Part B: (optional)
  120 mg ixekizumab given SC every 4 weeks. Subsequent to an amendment on May 2012, administration changed to 80 mg every 4 weeks through Week 236.
  Part C: (optional) 80 mg ixekizumab given SC every 4 weeks through approximately week 344.
  Interventions: Biological: Ixekizumab
- 80 mg Ixekizumab (Experimental): Part B: (optional)
  Subsequent to an amendment on May 2012, administration changed to 80 mg ixekizumab Q4W through Week 236.
  Part C: (optional) 80 mg ixekizumab given SC every 4 weeks through approximately week 344.
  Interventions: Biological: Ixekizumab

INTERVENTIONS:
Biological: Ixekizumab — Administered subcutaneously
  Other Names: LY2439821
Drug: Placebo — Administered subcutaneously
  Arms: Placebo

SUMMARY:
The primary purpose for this study is to help answer the following research questions

* The safety of ixekizumab (LY2439821) and any side effects that might be associated with it.
* Whether ixekizumab can help participants with Psoriasis.
* How much ixekizumab should be given to participants.

DETAILED DESCRIPTION:
The study is a Phase 2 study with 3 parts. Part A is a randomized, double-blind, placebo-controlled, parallel-group, dose-ranging design, Part B is an optional, open label extension design and Part C is an additional optional extension period with an open-label design(up to approximately 104 weeks). Approximately 125 participants will be randomized to 1 of 4 ixekizumab groups or to placebo (approximately 25 participants per group) in Part A. Participants will be evaluated for treatment efficacy and the primary endpoint will be evaluated at week 12. Between week 20 and week 32, participants with a less than 75% improvement in their Psoriasis Area and Severity Index (PASI) score compared to baseline will be eligible to begin Part B. Participants in Part B will receive subcutaneous (SC) injections of ixekizumab 120 milligrams (mg) every 4 weeks through week 236. Subsequent to an amendment on May 2012, administration changed to 80 mg every 4 weeks through Week 236. Participants in Part C may receive SC injections of ixekizumab 80 mg every 4 weeks for up to an additional 104 weeks through approximately week 340. Participants who complete Part A, Part B, and Part C will have a total study participation of approximately 344 weeks.

ELIGIBILITY:
Inclusion Criteria Common to Both Part A:

* Participant must have active plaque psoriasis covering at least 10% body surface area and a PASI score of at least 12 at screening and at randomization.
* Participant is a candidate for systemic therapy
* Participant has a Static Physician's Global Assessment (sPGA) score of at least 3 at screening and at randomization

Inclusion Criterion Specific to Part B

* Participant has completed the treatment period for part A (at least through week 20)

Inclusion Criterion Specific to Part C

* Participant has completed the treatment period for part B

Exclusion Criteria Common to Part A, B and C:

* Participant has pustular, erythrodermic and/or guttate forms of psoriasis
* Participant has had a clinically significant flare of psoriasis during the 12 weeks prior to study entry
* Participant has recently used any biologic agent/monoclonal antibody within the following washout periods: etanercept >28 days, infliximab or adalimumab >56 days, alefacept >60 days, ustekinumab >8 months, or any other biologic agent/monoclonal antibody >5 half-lives prior to baseline
* Participant has received systemic psoriasis therapy (such as psoralen and ultraviolet A [PUVA] light therapy, cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, azathioprine) or phototherapy (including ultraviolet B or self-treatment with tanning beds) within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to randomization (exception: class 6 [mild, such as desonide] or 7 [least potent, such as hydrocortisone] topical steroids will be permitted for use limited to the face, axilla, and/or genitalia)
* Participant has donated more than 500 mL of blood within the last month
* Participant has another serious disorder or illness
* Participant has suffered a serious bacterial infection (for example, pneumonia, and cellulitis) within the last 3 months
* Participant has a history of uncontrolled high blood pressure
* Participant has clinical laboratory test results at entry that are outside the normal reference range
* Participant is currently participating in or were discontinued within the last 30 days from another clinical trial involving an investigational drug
* Participant is a woman who is lactating or breast feeding
* If a participant is a woman and could become pregnant during this study, she must talk to the study doctor about the birth control that you will use to avoid getting pregnant during the study
* If a participant is post menopausal woman, she must be at least 45 years of age and have not menstruated for the last 12 months
* If a participant is a woman between 40-45 years of age, test negative for pregnancy, and have not menstruated during the last 12 months only, she must have an additional blood test to see if you can participate
* If the participant is male, he must agree to reduce the risk of female partner becoming pregnant during the study

Exclusion Criteria Specific to B:

* If a participant experienced a serious adverse event during Part A considered possibly related to ixekizumab
* If a participant experienced an adverse event during Part A that the study doctor believes continued ixekizumab treatment could cause harm to the participant.

Exclusion Criteria Specific to C:

* If a participant experienced a Serious Adverse Event during Part B considered possibly related to ixekizumab
* If a participant experienced an adverse event during Part B that the study doctor believes continued ixekizumab treatment could cause harm to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (31):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miramar, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newnan, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Skokie, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Dundee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jamaica, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Oswego, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., College Station, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hellerup

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Langley RG, Rich P, Menter A, Krueger G, Goldblum O, Dutronc Y, Zhu B, Wei H, Cameron GS, Heffernan MP. Improvement of scalp and nail lesions with ixekizumab in a phase 2 trial in patients with chronic plaque psoriasis. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1763-70. doi: 10.1111/jdv.12996. Epub 2015 Feb 18. PMID 25693783
- [Derived] Gordon KB, Leonardi CL, Lebwohl M, Blauvelt A, Cameron GS, Braun D, Erickson J, Heffernan M. A 52-week, open-label study of the efficacy and safety of ixekizumab, an anti-interleukin-17A monoclonal antibody, in patients with chronic plaque psoriasis. J Am Acad Dermatol. 2014 Dec;71(6):1176-82. doi: 10.1016/j.jaad.2014.07.048. Epub 2014 Sep 19. PMID 25242558
- [Derived] Leonardi C, Matheson R, Zachariae C, Cameron G, Li L, Edson-Heredia E, Braun D, Banerjee S. Anti-interleukin-17 monoclonal antibody ixekizumab in chronic plaque psoriasis. N Engl J Med. 2012 Mar 29;366(13):1190-9. doi: 10.1056/NEJMoa1109997. PMID 22455413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study has 3 parts:Part A is a randomized, double-blind, placebo-controlled, parallel-group, dose ranging design (approximately 20-40 weeks [wks]).Treatment durability (sustained efficacy off treatment) from Week 20 up to Week 32 was evaluated during Part A.
Pre-assignment Details: Part B is an optional extension period with an open-label design (approximately 240 weeks). Part C is an additional optional extension period with an open-label design(up to approximately 104 weeks).
Groups:
- Placebo: Part A:
  Placebo given on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 milligrams (mg) ixekizumab given subcutaneous (SC) every 4 weeks (Q4W). Subsequent to an amendment on May 2012, administration changed to 80 mg every 4 weeks through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through week 344.
- 10 mg Ixekizumab: Part A:
  10 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through week 344.
- 25 mg Ixekizumab: Part A:
  25 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through week 344.
- 75 mg Ixekizumab: Part A:
  75 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through week 344.
- 150 mg Ixekizumab: Part A:
  150 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  Administered 120 mg ixekizumab SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  Administered 80 mg ixekizumab SC Q4W through week 344.
- 120 mg/80 mg Total Ixekizumab: Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through week 344.
Period: Part A
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab | 120 mg/80 mg Total Ixekizumab
Started | 27 | 28 | 30 | 29 | 28 | 0 (120 mg and 80 mg ixekizumab were administered during Part B and C.)
Received at Least 1 Dose of Study Drug | 27 | 28 | 30 | 29 | 28 | 0 (120 mg and 80 mg ixekizumab were administered during Part B and C.)
Completed | 22 | 21 | 29 | 26 | 27 | 0 (120 mg and 80 mg ixekizumab were administered during Part B and C.)
Not Completed | 5 | 7 | 1 | 3 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Period: Part B and C
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab | 120 mg/80 mg Total Ixekizumab
Started | 0 (Placebo,10mg, 25mg,75mg and 150mg ixekizumab were administered during in Part A.) | 0 (Placebo,10mg, 25mg,75mg and 150mg ixekizumab were administered during in Part A.) | 0 (Placebo,10mg, 25mg,75mg and 150mg ixekizumab were administered during in Part A.) | 0 (Placebo,10mg, 25mg,75mg and 150mg ixekizumab were administered during in Part A.) | 0 (Placebo,10mg, 25mg,75mg and 150mg ixekizumab were administered during in Part A.) | 120 (80 and 120 mg ixekizumab were administered during Part B and C.)
Completed Part B (Week 240) | 0 | 0 | 0 | 0 | 0 | 74
Completed Part C | 0 | 0 | 0 | 0 | 0 | 0 (Part C was stopped once ixekizumab became available through marketing authorization.)
Post Treatment Safety Visits | 0 | 0 | 0 | 0 | 0 | 6 (Only participants with neutropenia entered the post treatment safety visits.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 (No participants completed the study as Part C was stopped.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 120
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 12
Not completed — Inclusion/Exclusion Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 10
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 66
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 16
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Part A:
  Placebo given on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  Part C: (optional)
  80 mg ixekizumab given SC Q4W through week 344.
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab | Total
Number analyzed (Participants) | 27 | 28 | 30 | 29 | 28 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12.76) | 47.65 (11.20) | 45.93 (14.53) | 46.37 (12.50) | 45.97 (13.00) | 46.19 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 12 | 10 | 14 | 61
  Male | 14 | 16 | 18 | 19 | 14 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 7 | 4 | 4 | 25
  Not Hispanic or Latino | 22 | 23 | 23 | 25 | 24 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 2 | 2 | 7
  White | 25 | 27 | 28 | 24 | 25 | 129
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 29 | 28 | 28 | 139
  Denmark | 0 | 1 | 1 | 1 | 0 | 3
Baseline in Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]).Overall scores range from 0 (no psoriasis) to 72(the most severe disease).
  units on a scale | 16.45 (5.26) | 19.18 (7.96) | 18.55 (4.94) | 17.20 (4.26) | 17.70 (6.21) | 17.83 (5.85)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index ≥75% (PASI 75) Improvement
Description: PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease).Participants achieving PASI 75 were defined as having an improvement of ≥75% in the PASI score compared to baseline.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline PASI assessment. Last Observation Carried Forward (LOCF) was used to impute missing post-baseline values.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Part A:
  Placebo given on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
- 10 mg Ixekizumab: Part A:
  10 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
- 25 mg Ixekizumab: Part A:
  25 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
- 75 mg Ixekizumab: Part A:
  75 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
- 150 mg Ixekizumab: Part A:
  150 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 26 | 28 | 30 | 29 | 28
percentage of participants | 7.7 | 28.6 | 76.7 | 82.8 | 82.1
Statistical Analysis 1: Comparison: Placebo vs 10 mg Ixekizumab; Test type: Superiority or Other; p = 0.079, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 25 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 75 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs 150 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Primary Outcome: Percentage of PASI Improvement From Baseline to 12 Week Endpoint
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease). Least squares (LS) mean values were calculated using mixed model repeated measures (MMRM) and controlled for baseline as a covariate, visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured.
Time Frame: Baseline to Week 12
Population: All randomized participants who received at least 1 dose of study drug, had at least 1 post-baseline PASI assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of improvement in PASI score
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 23 | 27 | 29 | 29 | 26
Percentage of improvement in PASI score | 16.22 [4.44 to 28.01] | 49.33 [38.25 to 60.41] | 78.48 [67.67 to 89.29] | 85.69 [74.87 to 96.50] | 87.12 [75.94 to 98.29]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 25 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 75 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo vs 150 mg Ixekizumab; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) Score of Cleared (0) or Minimal (1) With at Least a 2 Point Improvement" at Week 12
Description: The sPGA of psoriasis is scored on a 6-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 6 point severity scale (0 [clear] to 5 [severe]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the sPGA score and category (0=clear; 1=minimal; 2=mild; 3=moderate; 4=marked; 5 = severe). As defined by protocol, a responder is a participant who has a post-baseline sPGA score of '0' or a post-baseline score of '1' with at least a 2 point improvement from baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 26 | 28 | 30 | 29 | 28
percentage of participants | 7.7 | 25.0 | 70.0 | 72.4 | 71.4

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events Up to 20 Weeks
Description: Treatment-emergent adverse events (TEAEs) are events which were not present at baseline or pre-existing conditions at baseline that worsened in severity following the start of treatment. A summary of other non-serious Adverse Events (AEs), and all Serious Adverse Events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Up to 20 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 27 | 28 | 30 | 29 | 28
Participants | 17 | 21 | 21 | 17 | 13

5. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score at Week 16
Description: The HADS is a 14-item, participant self-reported scale that consists of an anxiety scale and a depression scale, each with 7 items. Items are rated on a 4-point Likert-type scale ranging from 0 (low level of anxiety or depression) to 3 (high level of anxiety or depression). Each subscale score ranges from 0 to 21 with higher scores indicating greater symptom severity. The classification is defined: 0-7 normal, 8-10 Borderline, 11-21 Abnormal. LS mean was calculated using the analysis of covariance (ANCOVA) model including treatment as fixed effect and baseline as covariate.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 25 | 28 | 29 | 29 | 28
units on a scale
  Anxiety | -0.86 (0.58) | -1.97 (0.55) | -2.10 (0.54) | -2.17 (0.54) | -2.81 (0.55)
  Depression | 0.17 (0.54) | -1.86 (0.51) | -1.75 (0.51) | -2.52 (0.51) | -2.01 (0.51)

6. Secondary Outcome: Change From Baseline in 16-Item Quick Inventory of Depressive Symptoms- Self Rated (QIDS-SR16) Total Score at Week 16
Description: The QIDS-SR16 is a self-administered, 16-item instrument in which a participant is asked to consider each statement as it relates to the way they have felt for the past 7 days. There is a 4-point scale for each item ranging from 0 (best) to 3 (worst). The 16 items are scored to give 9 individual depression domains (sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance [initial, middle and late insomnia or hypersomnia], decrease/increase in appetite/weight, and psychomotor agitation/retardation), which are summed to give a single score ranging from 0 to 27, with higher scores denoting greater symptom severity. The LS Mean (no multiplicity adjustments) are presented for each treatment versus placebo comparison at each visit and use an analysis of covariance (ANCOVA) model including baseline as a covariate and treatment as fixed effect in the model.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 24 | 27 | 26 | 27 | 25
units on a scale | -0.49 (0.56) | -1.56 (0.52) | -1.48 (0.53) | -2.13 (0.52) | -2.21 (0.54)

7. Secondary Outcome: Change From Baseline in Patient Global Assessment (PatGA) at Week 12
Description: The PatGA is a single-item self-reported instrument asking the participant to rate the severity of their psoriasis "today" by circling a number on the numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been). The LS Mean (no multiplicity adjustments) are presented for each treatment versus placebo comparison at each visit and use an analysis of covariance (ANCOVA) model including baseline as a covariate and treatment as fixed effect in the model.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 26 | 28 | 30 | 29 | 28
units on a scale | -0.6 (0.3) | -1.1 (0.3) | -2.3 (0.2) | -2.9 (0.3) | -2.5 (0.3)

8. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (VAS) at Week 12
Description: The pain VAS is a participant-administered single-item scale designed to measure current joint pain from psoriatic arthritis (PsA) using a 100- millimeter (mm) horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by placing a single mark on the horizontal 100-mm scale from 0mm (no pain) to 100 mm (pain as severe as you can imagine). A mixed effects model for repeated measures analysis was used. Least Squares (LS) Mean values were calculated using MMRM and were controlled for baseline as a covariate, visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline PASI assessment. Only participants with self-reported psoriatic arthritis at baseline were included in the analysis. Last Observation Carried Forward (LOCF) was used to impute missing post-baseline values.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter (mm)
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 4 | 7 | 11 | 8 | 8
millimeter (mm) | 3.87 [-20.90 to 28.64] | -4.32 [-23.05 to 14.41] | -19.36 [-34.31 to -4.40] | -21.24 [-37.89 to -4.58] | -34.24 [-51.83 to -16.66]

9. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-S) at Week 16
Description: MOS-S provides a concise assessment of important dimensions of sleep, including initiation, maintenance, respiratory problems, quantity, perceived adequacy, and somnolence during the past 4 weeks. Scoring based on 7 subscales: sleep disturbance, snoring, awakened short of breath or with headache, sleep adequacy, and somnolence (range:0-100,with higher scores for more impairment); sleep quantity (range:0-24), and optimal sleep (yes:1, no:0). Six(6) and 9 item index measures of sleep disturbance were constructed to provide composite scores. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range * 100); total score range: 0 to 100; higher score = higher scores indicate greater problems with the attribute.The LS Mean (no multiplicity adjustments) was calculated using an analysis of covariance (ANCOVA) model including baseline as a covariate and treatment as fixed effect in the model.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 25 | 28 | 29 | 29 | 28
units on a scale
  Sleep Problems Index I | -0.05 (2.61) | -5.35 (2.46) | -8.78 (2.42) | -7.97 (2.42) | -2.38 (2.47)
  Sleep Problems Index II | 0.21 (2.37) | -6.42 (2.24) | -9.23 (2.20) | -8.43 (2.20) | -2.48 (2.24)
  Sleep Adequacy | -2.83 (4.73) | 5.63 (4.47) | 11.35 (4.39) | 8.81 (4.39) | -0.41 (4.48)
  Sleep Disturbance | -1.47 (3.27) | -8.56 (3.10) | -10.02 (3.03) | -11.50 (3.04) | -4.67 (3.09)
  Sleep Somnolence | 1.12 (2.73) | -2.32 (2.58) | -7.14 (2.53) | -5.80 (2.53) | -0.76 (2.58)
  Snoring | -2.85 (4.22) | -0.47 (3.94) | 2.94 (3.88) | -3.24 (3.87) | -3.81 (3.94)
  Sleep Short of Breath/headache | 4.34 (3.10) | -5.45 (2.92) | -2.84 (2.87) | -2.65 (2.87) | -3.46 (2.91)

10. Secondary Outcome: Number of Participants Who Received Medical Care Measured by Medical Care Resource Utilization (PMRU))
Description: The PMRU is a 3-item participant-reported questionnaire on health care resource utilization due to psoriasis for physician/clinic visits, emergency room visits, and inpatient hospital admissions since the last study visit.
Time Frame: Week 16
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline PASI assessment.
Measure: Number; unit: participants
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 26 | 28 | 30 | 29 | 28
participants
  Week 16 - Office or Clinic(n=23,24,29,28,27) | 1 | 0 | 0 | 1 | 3
  Week 16 - Emergency Room(ER)(n=23, 24, 29, 28, 27) | 0 | 0 | 0 | 0 | 1
  Week 16 - Admitted thru ER (n=26,28,30,29,28) | 0 | 0 | 0 | 0 | 0
  Week 16 - Hospital Stay (n=26,28,30,29,28) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI Q) at Week 16
Description: The WPAI questionnaire has six questions to assess whether the participant was currently employed (Q1); how many hours from work were missed due to problems associated with psoriasis (Q2) or any other reason (Q3); hours actually worked (Q4); degree that psoriasis affected productivity while working (Q5); and degree that psoriasis affected regular activities (Q6) over the past 7 days. Four separate overall scores were calculated, Absenteeism (work time missed) = (Q2/(Q2+Q4))*100, Presenteeism(impairment at work/reduced on-the-job effectiveness) = (Q5/10) *100, Work productivity loss(overall work impairment /absenteeism plus presenteeism) = (Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))x(Q5/10)]) * 100 and Activity Impairment = (Q6/10) * 100. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity ( worse outcomes). The LS Mean was calculated using ANCOVA model including baseline as a covariate and treatment as fixed effect in the model.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 26 | 28 | 30 | 29 | 28
units on a scale
  Absenteeism (n=15,19,14,19,16) | -1.91 (1.88) | 0.71 (1.68) | -0.83 (1.94) | -2.64 (1.67) | -1.96 (1.82)
  Presenteeism (n=15,20,16,19,16) | -3.38 (3.99) | -0.99 (3.47) | -4.59 (3.87) | -14.48 (3.55) | -10.69 (3.90)
  Work productivity loss (n=15,19,14,19,16) | -3.65 (4.30) | 1.74 (3.82) | -4.65 (4.45) | -14.76 (3.82) | -11.12 (4.17)
  Activity Impairment (n=25,28,28,29,27) | -0.68 (4.19) | -9.76 (3.96) | -14.96 (3.95) | -12.81 (3.90) | -14.79 (4.03)

12. Secondary Outcome: Change From Baseline in Medical Outcomes Study Short-Form 36 (SF-36) - Physical Component Score (PCS) and Mental Component Score (MCS) at Week 16
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into the PCS and MCS scores. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. The recall period was the past 4 weeks. The LS Mean was calculated using ANCOVA model including baseline as a covariate and treatment as fixed effect in the model.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 25 | 28 | 28 | 29 | 28
units on a scale
  PCS | -1.22 (2.15) | 2.41 (2.03) | 1.95 (2.03) | 3.94 (2.00) | 5.72 (2.03)
  MCS | -0.56 (2.29) | 7.27 (2.19) | 5.16 (2.18) | 4.13 (2.13) | 4.15 (2.16)

13. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) in Participants With Nail Psoriasis at Week 12
Description: The NAPSI is physician-rated and quantifies the severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix and nail bed. Each finger nail is divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). Participant's fingers and toes were evaluated and the sum of the scores was added resulting in a range of 0 to 160; higher scores indicate greater severity. If an individual toe or finger assessment was missing (not done), the average of the remaining measured digits was imputed and added to the sum. If <50% of the toes or finger assessments were missing, the imputation was performed. If >50% of the assessments were missing, then the sum of the scores was left as missing. LS mean was calculated using MMRM with baseline score as covariate, visit, treatment and visit by treatment interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline PASI assessment. Only participants with baseline nail involvement were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 14 | 13 | 10 | 10 | 10
units on a scale | 2.21 [-5.17 to 9.58] | -4.85 [-12.82 to 3.12] | -3.65 [-12.73 to 5.43] | -15.89 [-24.98 to -6.81] | -19.91 [-29.00 to -10.83]

14. Secondary Outcome: Change From Baseline in Palmoplantar Psoriasis Severity Index (PPASI) in Participants With Palmoplantar Psoriasis at Week 12
Description: The PPASI is a physician-assessed composite score derived from the summed scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement. The PPASI score ranges from 0 to 72, with higher scores representing greater severity of palmoplantar psoriasis.LS mean was calculated using MMRM with baseline score as covariate, visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to symmetric.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline PASI assessment. Only participants with palmoplantar involvement were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 1 | 4 | 4 | 2 | 2
units on a scale | -1.0 [-10.3 to 8.3] | -6.4 [-12.3 to -0.5] | -4.6 [-10.3 to 1.2] | -3.4 [-11.5 to 4.8] | -12.8 [-20.9 to -4.7]

15. Secondary Outcome: Change From Baseline in Scalp Psoriasis Severity Index (PSSI) in Participants With Scalp Psoriasis at Week 12
Description: The PSSI is a physician-assessed composite score derived from the summed scores for erythema, induration, and desquamation multiplied by a score for the extent of scalp area involved. The PSSI score ranges from 0 to 72, with higher scores representing greater severity of scalp psoriasis.LS mean was calculated using MMRM with baseline score as covariate, visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline PASI assessment. Only participants with baseline scalp involvement were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 17 | 21 | 24 | 18 | 22
units on a scale | -7.3 [-11.2 to -3.5] | -10.2 [-13.9 to -6.6] | -15.8 [-19.2 to -12.4] | -15.0 [-18.9 to -11.0] | -17.2 [-20.8 to -13.7]

16. Secondary Outcome: Ixekizumab Systemic Clearance (CL) (Serum Concentrations of Ixekizumab From Baseline Through 32 Weeks)
Description: The population pharmacokinetic (PK) modeling value for systemic clearance was based on data from week 1 to week 32 for all participants in all ixekizumab treatment arms.
Time Frame: Week 1, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28 and Week 32
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (95% Confidence Interval); unit: liters per hour (L/hr)
Groups:
- All Participants (10mg, 25mg,75mg & 150 mg Ixekizumab): Part A:
  10 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  25 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  75 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
  150 mg ixekizumab given SC on weeks 0, 2, 4, 8, 12 and 16 for a total of six administrations.
Arm/Group | All Participants (10mg, 25mg,75mg & 150 mg Ixekizumab)
Number analyzed (Participants) | 115
liters per hour (L/hr) | 0.0177 [0.0160 to 0.0199]

17. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score Total Score at Week 16
Description: The DLQI is a 10-item, participant-administered dermatology-specific questionnaire that assess health related quality of life that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The DLQI items response categories are scored 0 (not relevant) to 3 (very much) with a total score range of 0 to 30; higher scores indicate poor quality of life and a 5-point change from baseline is considered clinically relevant. The LS Mean(no multiplicity adjustments) are presented for each treatment versus placebo comparison at each visit and use an analysis of covariance (ANCOVA) model including baseline as a covariate and treatment as fixed effect in the model.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 25 | 28 | 29 | 29 | 28
units on a scale | -1.24 (0.97) | -6.35 (0.92) | -6.59 (0.90) | -8.39 (0.90) | -8.17 (0.92)

18. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: PASI combines the extent of body surface involvement in 4 anatomical regions(head,trunk,arms,and legs).For each region the percent area of skin involved was estimated from 0(0%) to 6(90%-100%) and severity was estimated by clinical signs of erythema,induration and scaling with a scores range from 0(none) to 4(very severe).Each area is scored by itself and the scores were then combined for the final PASI.Final PASI calculated as:sum of severity parameters for each region*area score*weighing factor (head[0.1],upper limbs[0.2],trunk[0.3],lower limbs [0.4]).Overall scores range from 0(no psoriasis) to 72(most severe disease).The LS mean are presented for each treatment versus placebo comparison at each visit and use ANCOVA model including baseline PASI covariate and treatment as fixed effect in the model.Results at Week 12 are summarized as Improvement in PASI which is defined as a reduction in the PASI calculated score at a visit as compared to the score calculated at the baseline visit.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 26 | 28 | 30 | 29 | 28
units on a scale | 3.50 (1.21) | 8.20 (1.17) | 13.56 (1.12) | 14.99 (1.14) | 15.38 (1.16)

19. Secondary Outcome: Percentage of Participants Who Achieve a 75% Improvement in the Psoriasis Area and Severity Index (PASI 75)
Description: PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease). Participants achieving PASI 75 were defined as having an improvement of ≥75% in the PASI score compared to baseline.
Time Frame: Week 32
Population: All randomized participants who received at least 1 dose of study drug, completed study treatment in Part A, achieved PASI 75 at Week 20 and who were followed for treatment durability up to Week 32. Last Observation Carried Forward (LOCF) was used to impute missing post-baseline values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 6 | 22 | 23 | 23 | 23
percentage of participants | 0 | 50.0 | 59.1 | 56.5 | 82.6

20. Secondary Outcome: Percentage of PASI Improvement From Baseline Through 32 Weeks
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease). Improvement in PASI is defined as improvement in the PASI calculated score at a visit as compared to the score calculated at the baseline visit.
Time Frame: Baseline Through 32 Weeks
Population: All randomized participants who received at least 1 dose of study drug, completed study treatment in Part A, achieved PASI 75 at Week 20 and who were followed for treatment durability up to Week 32. Zero participants in the placebo arm had data.
Measure: Mean (Standard Deviation); unit: Percentage PASI improvement
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 0 | 4 | 16 | 18 | 21
Percentage PASI improvement |  | 80.55 (17.69) | 85.60 (12.74) | 85.16 (15.30) | 88.11 (11.35)

21. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) Score of Cleared (0) or Minimal (1) With at Least a 2 Point Improvement
Description: The sPGA of psoriasis is scored on a 6-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 6-point severity scale (0 [clear] to 5 [severe]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the sPGA score and category (0=clear; 1=minimal; 2=mild; 3=moderate; 4=marked; 5 = severe). As defined by protocol, a responder is a participant who has a post-baseline sPGA score of '0' or a post-baseline score of '1' with at least a 2 point improvement from baseline.
Time Frame: Week 32
Population: All randomized participants who received at least 1 dose of study drug, completed study treatment in Part A, achieved PASI 75 at Week 20 and who were followed for treatment durability up to Week 32. Last Observation Carried Forward (LOCF) was used to impute missing post-baseline values. Zero participants in the placebo arm had data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 0 | 6 | 22 | 23 | 23
percentage of participants |  | 33.3 | 45.5 | 47.8 | 65.2

22. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: Percentage of participants with treatment-emergent positive anti-ixekizumab antibodies was summarized by treatment group. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline through Week 20
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least one post-baseline antibody assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab
Number analyzed (Participants) | 25 | 24 | 30 | 29 | 27
percentage of participants | 4.0 | 54.2 | 40.0 | 17.2 | 22.2

23. Secondary Outcome: Percentage of Participants With Static Physician's Global Assessment (sPGA) of (0,1)
Description: as for outcome 21
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants who had PASI 75 response at Week 20.
Measure: Number; unit: percentage of participants
Groups:
- Total Ixekizumab (80 mg and 120 mg): Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
  During Part B of the study, participants were initially assigned to ixekizumab (LY2439821) 120 mg SC and were transitioned to ixekizumab 80 mg SC.
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 74
percentage of participants | 78.4

24. Secondary Outcome: Number of Treatment Emergent Adverse Events up to 344 Weeks
Description: as for outcome 4
Time Frame: Baseline Up to 344 Weeks
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 120
Participants | 105

25. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a 14-item, participant self-reported scale that consists of an anxiety scale and a depression scale, each with 7 items. Items are rated on a 4-point Likert-type scale ranging from 0 (low level of anxiety or depression) to 3 (high level of anxiety or depression). Each subscale score ranges from 0 to 21 with higher scores indicating greater symptom severity. The classification is defined: 0-7 normal, 8-10 Borderline, 11-21 Abnormal.
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants who had PASI 75 response at Week 20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 74
units on a scale
  Anxiety | -3.0 (3.4)
  Depression | -2.8 (3.0)

26. Secondary Outcome: Number of Participants With Patient's Global Assessment of Disease Activity (PatGA)
Description: The PatGA is a single-item self-reported instrument asking the participant to rate the severity of their psoriasis "today" by circling a number on the numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been).
Time Frame: Week 240
Population: All enrolled participants who had PASI 75 response at Week 20.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 74
Participants
  0(Clear) | 40
  1 | 26
  2 | 4
  3 | 2
  4 | 2
  5(Severe) | 0

27. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (VAS)
Description: The pain VAS is a participant-administered single-item scale designed to measure current joint pain from psoriatic arthritis (PsA) using a 100- millimeter (mm) horizontal VAS. Overall severity of participant's joint pain from PsA is indicated by placing a single mark on the horizontal 100-mm scale from 0mm (no pain) to 100 mm (pain as severe as you can imagine). A mixed effects model for repeated measures analysis was used.
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants with data available.
Measure: Mean (Standard Error); unit: Millimeters (mm)
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 24
Millimeters (mm) | -13.25 (32.34)

28. Secondary Outcome: Change From Baseline up to 240 Weeks in Nail Psoriasis Severity Index (NAPSI) in Participants With Nail Psoriasis
Description: The NAPSI is physician-rated and quantifies the severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix and nail bed. Each finger nail is divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). Participant's fingers and toes were evaluated and the sum of the scores was added resulting in a range of 0 to 160; higher scores indicate greater severity. If an individual toe or finger assessment was missing (not done), the average of the remaining measured digits was imputed and added to the sum. If <50% of the toes or finger assessments were missing, the imputation was performed. If >50% of the assessments were missing, then the sum of the scores was left as missing.
  Baseline is defined as the last available value prior to the first dose in Part A of the study.
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants with baseline nail psoriasis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 32
units on a scale | -33.62 (30.48)

29. Secondary Outcome: Change From Baseline up to 240 Weeks in Scalp Psoriasis Severity Index (PSSI) in Participants With Scalp Psoriasis
Description: The PSSI is a physician-assessed composite score derived from the summed scores for erythema, induration, and desquamation multiplied by a score for the extent of scalp area involved. The PSSI score ranges from 0 to 72, with higher scores representing greater severity of scalp psoriasis.
  Baseline is defined as the last available value prior to the first dose in Part A of the study.
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants with baseline scalp psoriasis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 56
units on a scale | -19.89 (13.68)

30. Secondary Outcome: Change From Baseline up to 240 Weeks in Palmoplantar Psoriasis Severity Index (PPASI) in Participants With Palmoplantar Psoriasis
Description: as for outcome 14
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants with baseline palmoplantar psoriasis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 4
units on a scale | -9.10 (7.59)

31. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index ≥75% (PASI 75) Improvement
Description: as for outcome 1
Time Frame: Week 240
Population: All enrolled participants who had PASI 75 response at Week 20.
Measure: Number; unit: percentage of participants
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 74
percentage of participants | 97.3

32. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI is a 10-item, participant-administered dermatology-specific questionnaire that assess health related quality of life that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The DLQI items response categories are scored 0 (not relevant) to 3 (very much) with a total score range of 0 to 30; higher scores indicate poor quality of life and a 5-point change from baseline is considered clinically relevant.
  Baseline is defined as the last available value prior to the first dose in Part A of the study.
Time Frame: Baseline Up to 240 Weeks
Population: All enrolled participants who had PASI 75 response at Week 20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Ixekizumab (80 mg and 120 mg)
Number analyzed (Participants) | 74
units on a scale | -9.2 (5.6)

ADVERSE EVENTS:
Description: Treatment durability refers to participants who had a PASI 75 response at Week 20 and remained in Part A of the study from Week 20-32 (treatment-free period). These participants moved to Part B of the study upon completion of Part A through Week 32 or upon loss of PASI75 response during the Part A treatment-free period.
Groups:
- Treatment Durability: Part A: Treatment durability/safety follow-up period:12 to 20 weeks.
- 120 mg and 80 mg Total Ixekizumab: Part B: (optional)
  120 mg ixekizumab given SC Q4W. Subsequent to an amendment on May 2012, administration changed to 80 mg Q4W through Week 236.
- Post Treatment Safety Visits: Participants who were followed due to neutropenia.
Arm/Group | Placebo | 10 mg Ixekizumab | 25 mg Ixekizumab | 75 mg Ixekizumab | 150 mg Ixekizumab | Treatment Durability | 120 mg and 80 mg Total Ixekizumab | Post Treatment Safety Visits
Serious Adverse Events (participants affected / at risk) | 1/27 | 1/28 | 1/30 | 0/29 | 0/28 | 1/74 | 24/120 | 0/6
Other Adverse Events (participants affected / at risk) | 13/27 | 15/28 | 12/30 | 10/29 | 11/28 | 11/74 | 82/120 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=27) | 10 mg Ixekizumab (N=28) | 25 mg Ixekizumab (N=30) | 75 mg Ixekizumab (N=29) | 150 mg Ixekizumab (N=28) | Treatment Durability (N=74) | 120 mg and 80 mg Total Ixekizumab (N=120) | Post Treatment Safety Visits (N=6)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/13 (0) | 0/12 (0) | 0/12 (0) | 0/10 (0) | 0/14 (0) | 0/33 (0) | 1/50 (1) | 0/4 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/13 (0) | 0/12 (0) | 0/12 (0) | 0/10 (0) | 0/14 (0) | 0/33 (0) | 1/50 (1) | 0/4 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/13 (1) | 0/12 (0) | 0/12 (0) | 0/10 (0) | 0/14 (0) | 0/33 (0) | 0/50 (0) | 0/4 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | 10 mg Ixekizumab (N=28) | 25 mg Ixekizumab (N=30) | 75 mg Ixekizumab (N=29) | 150 mg Ixekizumab (N=28) | Treatment Durability (N=74) | 120 mg and 80 mg Total Ixekizumab (N=120) | Post Treatment Safety Visits (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 9 (13) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (3) | 0 (0) | 4 (17) | 0 (0)
Peripheral swelling (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (16) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 9 (10) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 29 (57) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 17 (24) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 15 (21) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 13 (23) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (11) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (7) | 4 (11) | 1 (1) | 1 (1) | 3 (3) | 12 (20) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 8 (15) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 7 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days